CLINICAL TRIAL: NCT02003456
Title: Initial Human Validation of Simultaneous Dual-Tracer Cardiac PET Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Venkatesh L. Murthy, M.D., Ph.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00080193
Record Dates: First submitted 2013-11-04; First posted 2013-12-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Heart Disease; Myocardial Infarction
Keywords: positron emission tomography; rubidium; myocardial perfusion imaging; viability; FDG
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction | interventions — Rubidium-82; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac PET scan (Experimental): To evaluate methods that could allow the use of two radiotracers(rubidium-82/18F-fluorodeoxyglucose(FDG)and rubidium-82, that are used in cardiac positron emission tomography(PET)imaging scans to be performed at one time instead of the current method which involves being imaged at separate times, several hours apart.
  Interventions: Drug: Cardiac PET scan w/18F-Fluorodeoxyglucose and rubidium-82

INTERVENTIONS:
Drug: Cardiac PET scan w/18F-Fluorodeoxyglucose and rubidium-82 — Study subjects will undergo a Cardiac PET scan that will take approximately 20 minutes to complete. In addition to standard clinical rubidium-82/18F-fluorodeoxyglucose (FDG) PET imaging, during a separate imaging session, participants will be infused with a second dose of the radio-tracer rubidium-82 during FDG imaging scan that will take an additional 10 to 15 minutes to complete.
  Other Names: Positron emission tomography (PET Scan)

SUMMARY:
Positron emission tomography (PET) scans can be used to evaluate whether parts of the heart muscle are alive but receiving inadequate blood supply. This study involves the use of two radiotracers that will measure whether heart muscle cell are alive and quantify the blood supply to the heart muscle.

DETAILED DESCRIPTION:
Positron emission tomography (PET) scans can be used to evaluate whether parts of the heart muscle (myocardium) are alive but receiving inadequate blood supply. This information can be helpful in identifying the best course of treatment. This type of study involves the use of two radiotracers: rubidium-82 (to measure blood flow) and 18F-fluorodeoxyglucose or FDG (to measure whether heart muscle cells are alive). Currently, each of these radiotracers is imaged at separate times, several hours apart. The purpose of this study is to evaluate methods that could allow the entire study to be performed at one time.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Patients referred for clinically indicated positron emission tomography (PET) viability assessment with rubidium-82 rest perfusion imaging and 18F-fluorodeoxyglucose (FDG) metabolic imaging.

Exclusion Criteria:

1. Need for stress perfusion imaging
2. Claustrophobia which would prevent positron emission tomography (PET) imaging.
3. Inability to lie flat with arms positioned next to the head for approximately 20 minutes.
4. Clinical instability such as uncontrolled, potentially life threatening arrhythmias or heart failure requiring mechanical support or infusions of inotropic or vasopressor agents.
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Equivalence of Images from Rest Rubidium-82 Perfusion PET Obtained Separately versus Simultaneously | 2 years
  To establish that polar map images from rest rubidium-82 myocardial perfusion imaging performed prior to injection of 18F-fluorodeoxyglucose (FDG) as is routinely performed currently during clinical PET viability studies and rest rubidium-82 myocardial perfusion imaging performed simultaneously with FDG during the second half of an extended FDG imaging session are clinically equivalent.

SECONDARY OUTCOMES:
Equivalence of Quantitative Estimates of Global Myocardial Blood Flow using Rubidium-82 Perfusion PET Obtained Separately versus Simultaneously | 2 years
  To establish that quantitative estimates of global myocardial blood flow at rest determined from rubidium-82 myocardial perfusion imaging performed prior to injection of 18F-fluorodeoxyglucose (FDG) as is routinely performed currently during clinical PET viability studies and rest rubidium-82 myocardial perfusion imaging performed simultaneously with FDG during the second half of an extended FDG imaging session are clinically equivalent.
Equivalence of Images from FDG PET Obtained Separately versus Simultaneously | 2 Years
  To establish that FDG PET images obtained prior to injection of rubidium-82 and those obtained simultaneously with FDG during the second half of an extended FDG imaging session are clinically equivalent.

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh L. Murthy, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No